CLINICAL TRIAL: NCT05668169
Title: Family-centered Support Program for Caregivers of Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: wen yu Kuo, assistant professor (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, wen yu Kuo, assistant professor, assistant professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOST 110-2314-B-255-001 -
Record Dates: First submitted 2022-12-13; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Caregiver Burden
Keywords: family-centered intervention
MeSH Terms: conditions — Stroke; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: The family-centered support program included four components:
  (A) Stroke and rehabilitation education. (B) Problem-solving skills training. (C) Long-term care information support. (D) Instant messaging application-based 24-h peers-support group for caregivers.
Who Masked: Participant
Masking Description: To prevent contact between participants in the intervention and control groups, we allocated participants from the G ward to the intervention group and those from the H ward to the control group. Participants were not given information about the group allocations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-centered support program for caregivers of stroke survivors (Experimental): Participants receive usual hospital care and our intervention
  Interventions: Other: Family-centered support program for caregivers of stroke survivors
- No Intervention: Control group (No Intervention): Participants receive only usual hospital care

INTERVENTIONS:
Other: Family-centered support program for caregivers of stroke survivors — Once participants joined the family-centered support group, participants received 90-minute interventions, including an introduction to stroke and rehabilitation education, problem-solving skills training, and long-term care information. Investigators also invited participants to join the instant messaging application-based 24-h peer-support group for caregivers. On the second and fourth days after receiving the interventions, the researcher visited the participants to review and practice the content provided on the first day; each session was 30 to 40 minutes long. The researcher contacted the participants one week after participants joined the study to discuss their care difficulties or experiences and did so three times biweekly thereafter via the instant messaging application.
  Arms: Family-centered support program for caregivers of stroke survivors

SUMMARY:
The goal of this study is to evaluate the effect of a family-centered support program on the care burden, depressive symptoms, perceived social support, and quality of life of stroke survivor' caregivers and on care recipients' rehabilitation adherence and depressive symptoms.

DETAILED DESCRIPTION:
The family-centered support program included stroke and rehabilitation education, problem-solving skills training, long-term care information support, and instant messaging applications-based 24-h peers-support group for caregivers.

Investigators hypothesized that (1) Compared with those in the control group, caregivers who undergo a family-centered support program have lower care burdens, do not have a high risk of depression, and perceive better social support and quality of life; (2) Compared with those in the control group, care recipients in the family-centered support group have ideal rehabilitation adherence and are not at a high risk of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Caregivers:

   * Aged 20 years or older
   * Primarily responsible for caring for the stroke survivor in the hospital and after discharge.
2. Stroke survivors:

   * Diagnosed with moderate stroke (National Institute of Health Stroke Scale ≥5 or Modified Rank in Scale ≥3), including ischemic and hemorrhagic stroke, via computed tomography or magnetic resonance imaging within one month. admitted to the stroke unit at a medical center
   * Had a primary family caregiver.

Exclusion Criteria:

1. Caregivers:

   * Refusal to participate in the study
   * Unable to communicate, for example, non-Chinese speakers
   * Reported having been diagnosed with psychiatric illness (such as major depression) and undergoing treatment.
2. Stroke survivors:

   * Unstable vital signs
   * Terminal illness
   * Transfer to long-term care facilities after hospital discharge
   * Self-reported having been diagnosed with psychiatric illness (such as major depression) and undergoing treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | The outcome was assessed at baseline.
  Depressive symptoms were measured using the Taiwanese Depression Scale.The range of total scores is between 0~54, the scores higher than 19 indicated an increased risk of depression.
Caregiver care burden | The outcome was assessed at baseline.
  The caregiver strain index (CSI) was used to measure caregiver care burden. The range of total scores is between 0~13, the higher total scores indicated a higher care burden.
Perceived social support | The outcome was assessed at baseline.
  Medical Outcome Study Social Support Survey- Taiwanese version was used to measure the perceived social support for caregivers of stroke survivors. The range of total scores is between 19~95, and the higher full scores indicated a perception of better social support.
Caregivers' quality of life | The outcome was assessed at baseline.
  Taiwanese version of the World Health Organization Quality of Life BREF(WHOQOL-BREF) was used to measure caregivers' quality of life. The range of total scores is between 4~20, and the higher full scores indicated a better quality of life. WHOQOL-BREF was used to measure the quality of life of stroke survivors' caregivers.
Rehabilitation adherence | The outcome was assessed at baseline.
  A single item of rehabilitation adherence measurement was used to measure stroke Patients' rehabilitation adherence levels. The range of scores is between 1~5, and the highest scores indicated an optimal adherence level.
Change from baseline depressive symptoms at first month | The outcome was assessed at first month after inclusion.
  Depressive symptoms were measured using the Taiwanese Depression Scale.The range of total scores is between 0~54, the scores higher than 19 indicated an increased risk of depression.
Change from baseline caregiver care burden at first month | The outcome was assessed at first month after inclusion.
  The caregiver strain index (CSI) was used to measure caregiver care burden. The range of total scores is between 0~13, the higher total scores indicated a higher care burden.
Change from baseline perceived social support at first month | The outcome was assessed at first month after inclusion.
  Medical Outcome Study Social Support Survey- Taiwanese version was used to measure the perceived social support for caregivers of stroke survivors. The range of total scores is between 19~95, and the higher full scores indicated a perception of better social support.
Change from baseline caregivers' quality of life at first month | The outcome was assessed at first month after inclusion.
  Taiwanese version of the World Health Organization Quality of Life BREF(WHOQOL-BREF) was used to measure caregivers' quality of life. The range of total scores is between 4~20, and the higher full scores indicated a better quality of life.WHOQOL-BREF was used to measure the quality of life of stroke survivors' caregivers.
Change from baseline rehabilitation adherence at first month | The outcome was assessed at first month after inclusion.
  A single item of rehabilitation adherence measurement was used to measure stroke patients' rehabilitation adherence levels. The range of scores is between 1~5, and the highest scores indicated an optimal adherence level.
Change from baseline depressive symptoms at third month | The outcome was assessed at third after inclusion.
  Depressive symptoms were measured using the Taiwanese Depression Scale.The range of total scores is between 0~54, the scores higher than 19 indicated an increased risk of depression.
Change from baseline caregiver care burden at third month | The outcome was assessed at third after inclusion.
  The caregiver strain index (CSI) was used to measure caregiver care burden. The range of total scores is between 0~13, the higher total scores indicated a higher care burden.
Change from baseline perceived social support at third month | The outcome was assessed at third after inclusion.
  Medical Outcome Study Social Support Survey- Taiwanese version was used to measure the perceived social support for caregivers of stroke survivors. The range of total scores is between 19~95, and the higher full scores indicated a perception of better social support.
Change from baseline caregivers' quality of life at third month | The outcome was assessed at third after inclusion.
  Taiwanese version of the World Health Organization Quality of Life BREF (WHOQOL-BREF) was used to measure caregivers' quality of life. The range of total scores is between 4~20, and the higher full scores indicated a better quality of life. WHOQOL-BREF was used to measure the quality of life of stroke survivors' caregivers.
Change from baseline rehabilitation adherence at third month | The outcome was assessed at third after inclusion.
  A single item of rehabilitation adherence measurement was used to measure stroke patients' rehabilitation adherence levels. The range of scores is between 1~5, and the highest scores indicated an optimal adherence level.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No